CLINICAL TRIAL: NCT01952717
Title: A Multi-Reader Multi-Case Clinical Trial To Evaluate Diagnostic Accuracy of 3D Koning Breast CT Compared to 2D Diagnostic Mammography
Brief Title: PMA Required Pivotal Multi-reader Multi-case Reader Study
Status: Completed | Type: Observational
Sponsor: Koning Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: KBCT-006
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer Diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A pivotal multi-reader multi-case (MRMC) study to compare the diagnostic performance of 3D Koning Breast Computed Tomography (KBCT) to that of 2D Diagnostic Mammography to support the Pre-market Approval (PMA) of KBCT by the US Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
This study will be conducted according to US and international standards of Good Clinical Practice (FDA regulations 21 CFR 11, 50, 56, and 812 and FDA guidance E6). Applicable government regulations and Medical University of South Carolina research policies and procedures will also be followed.

The goal of the study is to evaluate if 3D KBCT can improve the clinical performance of diagnostic workup for breast cancer detection and diagnosis compared to 2D Diagnostic Mammography.

This study will involve 18 readers reading and scoring the conventional 2D diagnostic mammograms and the 3D KBCT images of 236 cases. Each reader will undergo one day of training prior to beginning the reader study. The reader study will be broken up into one three-day reading session (includes training day) and three two-day reading sessions with a washout period of at least four weeks in between sessions.

The 2D diagnostic mammograms include standard 2-view mammograms and any additional diagnostic views. The ROC curves will be constructed for 2D Diagnostic Mammography, 3D KBCT plus Standard 2-view Mammography (CC and MLO) (screening or diagnostic), and 3D KBCT. The area under the ROC curve (AUC) will be compared. The clinical decision regarding biopsy will also be evaluated by estimating the sensitivity and specificity of 2D Diagnostic Mammography, 3D KBCT plus Standard 2-view Mammography (CC and MLO), and 3D KBCT.

This study, including the training of the participating radiologists, will be conducted at the Department of Radiology at Medical University of South Carolina.

ELIGIBILITY:
Inclusion Criteria:

- At least 40 or 35 years of age of any ethnicity Had a routine mammogram, read as BI-RADS® 3 Have a palpable abnormality detected by Breast Self Exam (BSE), or Clinical Breast Exam (CBE) or have a non-palpable abnormality detected by an imaging modality After diagnostic work-up are categorized as BI-RADS® 4 or 5. Are scheduled for biopsy either by large gauge needle biopsy or excisional biopsy.

Will undergo study imaging prior to biopsy and within four weeks of diagnostic work-up Is able to provide informed consent

Exclusion Criteria:

- Pregnancy Lactation Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker Subjects who are unable to tolerate study constraints Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to) Treatment for enlarged thymus gland as an infant Irradiation for benign breast conditions, including breast inflammation after giving birth Treatment for Hodgkins disease Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to) Tuberculosis Severe scoliosis

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve 18 readers reading and scoring the conventional 2D diagnostic mammograms and the 3D KBCT images of 236 cases.
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver Operating Characteristics Curve (AUC) | one three-day reading session (includes training day) and three two-day reading sessions with a washout period of at least four weeks in between sessions
  The 2D diagnostic mammograms include standard 2-view mammograms and any additional diagnostic views. The ROC curves will be constructed for 2D Diagnostic Mammography, 3D KBCT plus Standard 2-view Mammography (CC and MLO) (screening or diagnostic), and 3D KBCT. The area under the ROC curve (AUC) will be compared.